CLINICAL TRIAL: NCT05050279
Title: A Phase 1 Clinical Trial to Evaluate QTcF Prolongation and Proarrhythmic Potential of the Non Antiarrhythmic Drug Delgocitinib Following Oral Administration in Healthy Subjects
Brief Title: A Trial to Evaluate the Effect of Delgocitinib on the Heart Rhythm of Healthy People
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: LP0133-1409
Record Dates: First submitted 2021-07-05; First posted 2021-09-20 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2022-01

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — delgocitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Placebo (Placebo Comparator): Delgocitinib placebo capsule
  Interventions: Drug: Placebo capsule
- Active dose 1 (Experimental): Delgocitinib capsule (Dose 1)
  Interventions: Drug: Delgocitinib capsule
- Active dose 2 (Experimental): Delgocitinib capsule (Dose 2)
  Interventions: Drug: Delgocitinib capsule
- Active dose 3 (Experimental): Delgocitinib capsule (Dose 3)
  Interventions: Drug: Delgocitinib capsule
- Active dose 4 (Experimental): Delgocitinib capsule (Dose 4)
  Interventions: Drug: Delgocitinib capsule

INTERVENTIONS:
Drug: Delgocitinib capsule — oral capsule
  Arms: Active dose 1; Active dose 2; Active dose 3; Active dose 4
Drug: Placebo capsule — oral capsule
  Arms: Placebo

SUMMARY:
The purpose of this trial is to investigate the effects of delgocitinib, taken as a capsule, on the heart rhythms of healthy people, compared to a placebo.

DETAILED DESCRIPTION:
The trial will be performed in two parts.

* Part 1: Group 1 (dose 1 or placebo) and Group 2 (dose 2 or placebo)
* Part 2: Group 3 (dose 3 or placebo) and Group 4 (dose 4 or placebo)

The doses in Part 2 may be adjusted depending on the results of Part 1.

Participants will be screened within 28 days of their dose. Participants will stay in the clinic from Day -1 to Day 2 (1 day postdose) and will be dosed on Day 1. A follow up phone call will take place 2 week (±2 days) after dosing.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index of ≥18.0 and <30.0 kg/m2.
* In good health, as judged by the investigator based on: medical history, physical examination, vital sign assessment, clinical laboratory evaluations .
* ECG without any clinically relevant abnormal findings at both screening and baseline
* No history of additional risk factors for torsades de pointes (for example, heart failure, hypokalaemia, family history of long QT syndrome).
* Female subjects of childbearing potential and male subjects with a female partner of childbearing potential must be willing to use highlly effective methods of contraception.

Exclusion Criteria:

* Any disorder which is not stable and could:

  * Affect the safety of the subject throughout the trial.
  * Influence the findings of the trial.
  * Impede the subject's ability to complete the trial.
* Use of any medication known to prolong the QT/QTc interval within 3 months or 5 half-lives of the drug, whichever is longer, prior to randomisation.
* Any medications, including St. John's wort, known to chronically alter drug absorption or elimination processes within 30 days prior to dosing.
* Current use of combined hormone contraceptives or combined hormonal replacement therapy.
* Subjects who have smoked (use of any type of tobacco and nicotine containing products) within the last 3 months prior to screening.
* History of chronic alcohol or drug abuse within 12 months prior to screening.
* Receipt of any vaccine approved for SARS-CoV-2 within 4 weeks prior to baseline and/or 2 weeks after dose.
* Receipt of live, attenuated vaccines within 4 weeks prior to baseline.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2021-09-29 (Actual); Primary Completion 2022-01-04 (Actual); Study Completion 2022-01-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline QTcF (ΔQTcF) | predose to 24 hours postdose
  Replicate electrocardiograms (ECGs) (10 ECG replicates) for the determination of ΔQTc interval will be extracted from the continuous digital 12-lead ECG recording

SECONDARY OUTCOMES:
Placebo-corrected change from baseline QTcF (ΔΔQTcF) | predose to 24 hours postdose
  Replicate electrocardiograms (ECGs) (10 ECG replicates) for the determination of ΔΔQTc interval will be extracted from the continuous digital 12-lead ECG recording
Change from baseline of Heart Rate (ΔHR) | predose to 24 hours postdose
  Replicate electrocardiograms (ECGs) (10 ECG replicates) for the determination of ΔHR interval will be extracted from the continuous digital 12-lead ECG recording
Placebo-corrected, change from baseline of Heart Rate (ΔΔHR) | predose to 24 hours postdose
  Replicate electrocardiograms (ECGs) (10 ECG replicates) for the determination of ΔΔHR interval will be extracted from the continuous digital 12-lead ECG recording
Change from baseline of Pulse Rate (ΔPR) | predose to 24 hourse postdose
  Measurement of PR will be performed manually from electrocardiograms (ECGs).
Placebo-corrected, change from baseline of Pulse Rate (ΔΔPR) | predose to 24 hours postdose
  Measurement of PR will be performed manually from electrocardiograms (ECGs).
Change from baseline of QRS interval (ΔQRS) | predose to 24 hours postdose
  Measurement of QRS will be performed manually from electrocardiograms (ECGs).
Placebo-corrected, change from baseline of QRS interval (ΔΔQRS) | predose to 24 hours postdose
  Measurement of QRS will be performed manually from electrocardiograms (ECGs).
Frequency of treatment emergent changes in T-wave morphology. | predose to 24 hours postdose
  Measurement of T-wave morphology will be performed manually
Frequency of treatment emergent changes in U-waves presence | predose to 24 hours postdose
  Measurement of U-waves presence will be performed manually
Categorical outliers for QTcF, HR, PR interval, and QRS duration. | predose to 24 hours post-dose
  Analysis perfomed for changes in categorical outlines based on treatment emergent adverse events.
Number of treatment emergent adverse events | dosing to day 15

CONTACTS AND LOCATIONS:
Overall Officials: Medical Expert, Study Director — LEO Pharma
Locations (1):
- Labcorp Clinical Research Unit (CRU) Ltd, Springfield House, Hyde Street,, Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Thaci D, Gooderham M, Lovato P, Madsen DE, Soehoel A, Bissonnette R. Systemic exposure and bioavailability of delgocitinib cream in adults with moderate to severe Chronic Hand Eczema. J Eur Acad Dermatol Venereol. 2025 Sep;39(9):1612-1621. doi: 10.1111/jdv.20777. Epub 2025 Jun 17. PMID 40525591